CLINICAL TRIAL: NCT04779294
Title: The Oslo Stan vs Lactate Observational Study, an Observational Study Were we Compare the Clinical Performance of Two Adjunctive Methods to CTG in Intrapartum Fetal Monitoring
Brief Title: The Oslo Stan vs Lactate Observational Study
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: Haukeland University Hospital (Other)
Responsible Party: Principal Investigator, Anne Flem Jacobsen, Senior Consultant, dpt of Obstetrics, Prof II University of Oslo, Oslo University Hospital
Other Study IDs: 2017/1561
Record Dates: First submitted 2019-12-12; First posted 2021-03-03 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: Fetal Monitoring
Keywords: CTG; Fetal blood sampling - Lactate; ST waveform analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fetus in labour at risk of acedimia: The Group of patients studied are fetuses in labour at risk of hypoxia with internal fetal monitoring and scalp lactate bloodsamples ( standard monitoring).
  Interventions: Diagnostic Test: STAN ( St wave analysis) and fetal blood sample-lactate
- Fetus in labour at risk of acedemia with STAN analysis: Same group of fetuses in labour at risk of hypoxia with internal fetal monitoring and STAN analysis(ST waveform analysis of the fetal electrocardiogram, opened after study inclusion finished)
  Interventions: Diagnostic Test: STAN ( St wave analysis) and fetal blood sample-lactate

INTERVENTIONS:
Diagnostic Test: STAN ( St wave analysis) and fetal blood sample-lactate — The CTG will be analysed by an expert group additional to the standard procedure that have been done in Labour already. The STAN analysis will be decrypted/ demasked anonymously by the Company producing these machines.

SUMMARY:
The main aim of the study is to compare the clinical performance of two adjunctive methods to CTG in intrapartum fetal monitoring: FBS with measurement of scalp lactate and ST analysis of the fetal ECG.

DETAILED DESCRIPTION:
We use Lactate as a standard adjunctive method in our hospital but we have STAN software available ( is demasked) in our CTG monitors. We will include all women in labour with an intern scalp monitoring and analyse the CTG, the lactate samples and the STAN signals in the same patient and

* Study the relationship between the decision-to-delivery interval and neonatal morbidity in deliveries monitored by scalp lactate measurement
* Compare the diagnostic capability of both methods to identify fetuses at risk of hypoxia
* Compare the false negative alerts from both methods
* Explore the temporal and quantitative relation between fetal lactate metabolism and ST interval changes of the fetal ECG

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Cephalic presentation
* Gestational age ≥36+0 weeks at delivery
* Presence of antpartum or intrapartum risk factors for fetal hypoxia according to Norwegian guidelines and therefore indication for electronic fetal monitoring with scalp electrode .

Exclusion Criteria:

* Multiple pregnancies
* Breech presentation
* Gestational age < 36+0 weeks
* Contraindications for placement of a scalp electrode (HIV or HBV or HCV pos)

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only women who are pregnant
Study Population: Women in labour who are monitored with CTG and FBS scalp lactate. CTG monitoring is achieved by an internal scalp electrode combined with a pressure-sensitive external contraction transducer. FBS is performed at the decision of the obstetrician. Capillary blood is obtained from the fetal head and analyzed with a bed-side test (Lactate Pro). The monitoring procedures described above are identical with the current clinical routine at the department.
  The department utilizes S31 fetal monitors (Neoventa Medical AB©, Sweden), which are equipped with the hard and software tool for ST analysis. Once the scalp electrode is attached, ST analysis will be performed and recorded continuously. ST information is blinded in labor, i.e. clinical management will only be based on CTG and FBS if indicated.
Sampling Method: Probability Sample
Enrollment: 694 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Is fetal hypoxia (defined as arterial umbilical cord pH < 7,1 postpartum) superiorly identified by fetal scalp blood sampling (lactate) or ST analysis of fetal ECG | 2019-2022
  1. Compare the diagnostic capability of both methods to identify fetuses at risk of hypoxia (i.e.umbilical artery blood pH ≤7.1)
  2. Compare FBS lactate with STAN in order to identify the superior method to avoid cord-blood acidosis at birth (i.e.umbilical artery blood pH >7.1)
  3. Compare the true negative alerts from both methods, specificity
Is cord blood acidosis, measured as pH in the umbilical artery postpartum affected by the "Decision-to-delivery interval" measured in minutes from Lactate warning until delivery. | 2019-2022
  To assess the effect of increasing time interval from the objective warning of intrapartum fetal hypoxia with fetal scalp lactate ≥ 4.8mmol/l to the end of operative delivery on the percentage of moderate cord-blood acidosis at birth (i.e., umbilical artery blood pH ≤ 7.1)

CONTACTS AND LOCATIONS:
Overall Officials: Jacobsen F Anne Flem, MD, PhD, Study Director — OUH
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berge MB, Kessler J, Staff AC, Jacobsen AF. The diagnostic accuracy of different fetal blood sample lactate cutoffs in labor, utilizing the StatStrip Xpress(R) lactate-meter: A population-based observational study. Acta Obstet Gynecol Scand. 2025 Aug;104(8):1496-1504. doi: 10.1111/aogs.15140. Epub 2025 Apr 30. PMID 40304212
- [Derived] Berge MB, Jacobsen AF, Yli BM, Staff AC, Gunnes N, Falk RS, Helgadottir LB, Kessler J. A direct comparison of the diagnostic accuracy of ST segment analysis (STAN) and fetal scalp blood sample lactate: A population-based observational study. Eur J Obstet Gynecol Reprod Biol. 2025 Apr 17;308:147-152. doi: 10.1016/j.ejogrb.2025.03.002. Epub 2025 Mar 3. PMID 40054097
- [Derived] Berge MB, Kessler J, Yli BM, Staff AC, Gunnes N, Jacobsen AF. Neonatal outcomes associated with time from a high fetal blood lactate concentration to operative delivery. Acta Obstet Gynecol Scand. 2023 Aug;102(8):1106-1114. doi: 10.1111/aogs.14597. Epub 2023 Jun 7. PMID 37287317